CLINICAL TRIAL: NCT00773617
Title: Integrative Cognitive Affective Therapy for Bulimia Nervosa (ICAT)
Brief Title: Testing an Alternative Therapy for Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH077571 (NIH); R34MH077571 (NIH); 5R34MH077571-02 (NIH)
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2013-04

CONDITIONS: Eating Disorders
Keywords: Bulimia Nervosa; Treatment Efficacy; Integrative Cognitive Affective Therapy; Cognitive Behavior Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Integrative cognitive affective therapy (ICAT)
  Interventions: Behavioral: ICAT
- 2 (Active Comparator): Cognitive behavioral therapy (CBT)
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: ICAT — ICAT is a new manual-based psychotherapy treatment for bulimia nervosa (BN) that focuses on emotions and bulimic behavior.
  Arms: 1
Behavioral: CBT — CBT is a highly structured, manual-based psychotherapy that has been shown to be effective in the treatment of BN. CBT focuses on cognitions and bulimic behavior.
  Arms: 2

SUMMARY:
This study will compare a new method of treatment for bulimia nervosa (ICAT), integrative cognitive-affective therapy, to the current standard method of treatment, cognitive behavioral therapy (CBT).

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a disorder characterized by binge eating and compensatory behaviors, such as self-induced vomiting or laxative abuse. It affects 1% to 2% of adolescents and young women, and occurs more rarely in men. People who suffer from BN are also more likely to suffer from other psychiatric disorders, such as anxiety disorders, mood disorders, substance abuse disorders, and personality disorders-those categorized as Axis II in the DSM IV.

Integrative cognitive-affective therapy (ICAT) is a new treatment developed as an alternative to cognitive behavioral therapy (CBT) for treating people with BN. CBT is the standard treatment for BN. ICAT uses some elements from CBT and some elements from therapies used to treat other disorders. Some elements of ICAT are also used to treat substance abuse disorders, depression, and personality disorders. This study will compare the effectiveness of ICAT and CBT in treating BN.

Participants in this study, who must have BN symptoms, will be randomly assigned to receive either CBT or ICAT treatment. Participation in this study will last 18 weeks for participants assigned to receive CBT and 16 weeks for participants assigned to receive ICAT. Both treatments will consist of 20 individual therapy sessions lasting 50 minutes. Additionally, participants receiving ICAT will receive personal digital assistant (PDA) devices installed with therapeutic modules. Use of these modules will be unlimited during the period of ICAT treatment and will be recorded at study visits. Over the course of 2 screening visits, participants will complete questionnaires, undergo clinical interviews, and go through a medical screening that involves a blood test of electrolytes and a urine test for pregnancy. Each screening visit will take 2 to 3 hours. At the end of treatment and 4 months after treatment completion, participants will undergo 2 assessments, both of which will include 2 hours of interviews and questionnaires. During these assessments researchers will evaluate weight; eating behavior; and associated problems with mood, anxiety, obsessive-compulsive symptoms, self-concept, social adjustment, and other areas of psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Bulimia nervosa, as defined by DSM-IV, or bulimic symptoms, as defined as purging episodes (with objective or subjective binge eating) that occur at least once per week for the past 3 months

Exclusion Criteria:

* Past or current diagnosis of psychosis or bipolar disorder
* Inability to read English
* Medical instability, including electrolyte abnormalities
* Psychotherapy or pharmacotherapy initiated within 6 weeks of study entry
* Pregnant or lactating
* Drug or alcohol dependence in the past 6 months or drug or alcohol abuse in the past 6 weeks
* Severe cognitive impairment or mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Percent reduction in binging or purging frequency as defined by symptom recall (SR) | Measured at baseline, weekly intervals throughout the duration of therapy, end of treatment, and 32-week follow-up
Percent reduction in binging or purging frequency, as defined by the Eating Disorders Examination (EDE) | Measured at baseline, end of treatment, and 32-week follow-up

SECONDARY OUTCOMES:
Reduction in depression, as defined by the Beck Depression Inventory (BDI) | Measured at baseline, therapy session eight, end of treatment, and 32-week follow-up
Reduction in anxiety as defined by the State-Trait Anxiety Inventory (STAI) | Measured at baseline, therapy session eight, end of treatment, and 32-week follow-up
Abstinence from binging and purging behavior, as defined by SR and EDE | Measured at the end of treatment and 32-week follow-up
Study retention rates | Measured weekly throughout treatment
Patient and therapist satisfaction, as defined by the Treatment Acceptability, Feasibility and Satisfaction Scale (TAFSQ) | Measured at therapy session two, therapy session eight, end of treatment, and 32-week follow-up
Self-esteem, as defined by the Rosenberg Self Esteem Questionnaire (RSEQ) | Measured at baseline, therapy session eight, end of treatment, and 32-week follow-up
Self-discrepancy, as defined by the Selves Interview | Measured at baseline, end of treatment, and at 32-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Wonderlich, PhD, Principal Investigator — Neuropsychiatric Research Institute, University of North Dakota
Locations (2):
- United States (2):
  - University of Minnesota Eating Disorders Research Program, Minneapolis, Minnesota
  - Neuropsychiatric Research Institute, Fargo, North Dakota

REFERENCES:
- [Derived] Peterson CB, Berg KC, Crosby RD, Lavender JM, Accurso EC, Ciao AC, Smith TL, Klein M, Mitchell JE, Crow SJ, Wonderlich SA. The effects of psychotherapy treatment on outcome in bulimia nervosa: Examining indirect effects through emotion regulation, self-directed behavior, and self-discrepancy within the mediation model. Int J Eat Disord. 2017 Jun;50(6):636-647. doi: 10.1002/eat.22669. Epub 2017 Jan 24. PMID 28117906
- [Derived] Haynos AF, Pearson CM, Utzinger LM, Wonderlich SA, Crosby RD, Mitchell JE, Crow SJ, Peterson CB. Empirically derived personality subtyping for predicting clinical symptoms and treatment response in bulimia nervosa. Int J Eat Disord. 2017 May;50(5):506-514. doi: 10.1002/eat.22622. Epub 2016 Sep 9. PMID 27611235
- [Derived] Accurso EC, Wonderlich SA, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ, Berg KC, Peterson CB. Predictors and moderators of treatment outcome in a randomized clinical trial for adults with symptoms of bulimia nervosa. J Consult Clin Psychol. 2016 Feb;84(2):178-84. doi: 10.1037/ccp0000073. Epub 2015 Dec 21. PMID 26689304
- [Derived] Accurso EC, Fitzsimmons-Craft EE, Ciao A, Cao L, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ, Wonderlich SA, Peterson CB. Therapeutic alliance in a randomized clinical trial for bulimia nervosa. J Consult Clin Psychol. 2015 Jun;83(3):637-42. doi: 10.1037/ccp0000021. Epub 2015 Apr 20. PMID 25894667
- [Derived] Wonderlich SA, Peterson CB, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ. A randomized controlled comparison of integrative cognitive-affective therapy (ICAT) and enhanced cognitive-behavioral therapy (CBT-E) for bulimia nervosa. Psychol Med. 2014 Feb;44(3):543-53. doi: 10.1017/S0033291713001098. Epub 2013 May 23. PMID 23701891